CLINICAL TRIAL: NCT00329394
Title: Study of the Efficacity of the Systemic Ketamine for the Improvement of Post-Operative Analgesia After ORL Carcinological Surgery at the Alcohol-Dependent Patient.
Brief Title: Systemic Ketamine for the Improvement of Post-Operative Analgesia at the Alcohol-Dependent Patient
Status: Suspended | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Dr Nicolas RASCOL, CHU Clermont-Ferrand
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CHU63-008
Record Dates: First submitted 2006-05-23; First posted 2006-05-24 (Estimated); Last update posted 2008-10-08 (Estimated); Status verified 2008-10

CONDITIONS: Alcoholic Patient; Carcinological Surgery ORL
Keywords: Ketamine; Analgesia; Alcool-dependent; carcinological surgery
MeSH Terms: conditions — Agnosia | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: ketamine — Evaluate the analgesic effectiveness of the systemic ketamine on the control of pain in the alcohol-dependent patient

SUMMARY:
The principal objective is to evaluate the analgesic effectiveness of the systemic ketamine on the control of the pain (average consumption of morphine at 48 hours) at the alcool-dependent patient, in carcinological surgery ORL. The effect coanalgesic is found for low dose of ketamine and action anti NMDA seems to have a stabilizing effect on this particular type of patient. This imbalance of the receivers, with a greater number of r-NMDA among these patients would involve it a better analgesic effectiveness and less effects dysphoric, to see an improvement on the syndrome of weaning. The secondary objectives evaluate the pain, the ground (dependence with alcohol), the first request analgesic, the tolerance and the signs psychic (syndrome of weaning...) and the satisfaction of the patient.

DETAILED DESCRIPTION:
The principal objective is to evaluate the analgesic effectiveness of the systemic ketamine on the control of the pain (average consumption of morphine at 48 hours) at the alcool-dependent patient, in carcinological surgery ORL. The effect coanalgesic is found for low dose of ketamine and action anti NMDA seems to have a stabilizing effect on this particular type of patient. This imbalance of the receivers, with a greater number of r-NMDA among these patients would involve it a better analgesic effectiveness and less effects dysphoric, to see an improvement on the syndrome of weaning. The secondary objectives evaluate the pain, the ground (dependence with alcohol), the first request analgesic, the tolerance and the signs psychic (syndrome of weaning...) and the satisfaction of the patient.

ELIGIBILITY:
Inclusion Criteria:

* patient alcohol-dependent having to undergo a carcinological surgery ORL with tracheotomy or tracheostomy, ASA 1-3

Exclusion Criteria:

* refusal of the patient
* counter-indications with the treatments,
* urgency
* the specific clinical context (final neoplasy, reanimation)
* the treatments for chronic pain containing morphinic

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2006-04; Primary Completion 2008-09 (Estimated); Study Completion 2008-09 (Estimated)

PRIMARY OUTCOMES:
Morphine consumption at 48 hours | at 48 hours

SECONDARY OUTCOMES:
pain | pain
the ground (dependence with alcohol) | dependence with alcohol
the first request analgesic | the first request analgesic
the tolerance and the signs psychic (syndrome of weaning...) | the tolerance and the signs psychic
and the satisfaction of the patient | the satisfaction of the patient

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Rascol, Dr, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Clermont-Ferrand University Hospital, Clermont-Ferrand, France

REFERENCES:
- [Background] Elia N, Tramer MR. Ketamine and postoperative pain--a quantitative systematic review of randomised trials. Pain. 2005 Jan;113(1-2):61-70. doi: 10.1016/j.pain.2004.09.036. PMID 15621365
- [Background] Petrakis IL, Limoncelli D, Gueorguieva R, Jatlow P, Boutros NN, Trevisan L, Gelernter J, Krystal JH. Altered NMDA glutamate receptor antagonist response in individuals with a family vulnerability to alcoholism. Am J Psychiatry. 2004 Oct;161(10):1776-82. doi: 10.1176/ajp.161.10.1776. PMID 15465973